CLINICAL TRIAL: NCT07397585
Title: stereOtactic Body RadIothErapy for exTracranial oligomeTastAtic Breast Cancer: Multi Institutional Retrospective Database
Acronym: ORIETTA
Status: Recruiting | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: RT/OSS - 001/2025
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer; Oligometastasis
Keywords: breast cancer; oligometastasis; radiotherapy; SBRT
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TREATMENT SBRT: patients who have been treated with stereotactic radiotherapy to oligometastatic sites

SUMMARY:
Oligometastatic breast cancer is a condition in which breast cancer has spread to a small number of other parts of the body. Patients with this type of disease may live longer than those with more widespread metastases. In addition to standard treatments that act on the whole body, such as chemotherapy or hormonal therapy, these patients might also benefit from local treatments that directly target the cancer spots. One of these local treatments is stereotactic body radiotherapy (SBRT), a non-invasive radiation treatment that delivers high doses of radiation in a few sessions. In the past, most of the evidence about the benefit of local treatments came from surgery. More recently, there has been growing interest in SBRT because it does not require surgery. However, the results of studies so far have not been consistent.The goal of this multicenter retrospective study is to better understand whether SBRT can improve disease control and survival in patients with breast cancer that has spread to a limited number of sites outside the brain.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years
* Histological diagnosis of breast cancer
* Oligometastatic or oligoprogressive metastatic breast cancer
* SBRT delivered to a minimum dose of 50Gy EQD2 (αβ 10 Gy),in a maximum of 12 fractions as per Oligocare definition
* Ability to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with Oligometastatic or oligoprogressive metastatic breast cancer treated with SBRT
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
progression free survival | from January 2010 to December 2023
  years of survival without disease progression assessed by imaging

SECONDARY OUTCOMES:
Local Control | from January 2010 to December 2023
  time between treatment and disease recurrence assessed by imaging
overall survival | From January 2010 to December 2023
  the time from diagnosis or initiation of treatment until death from any cause
acute and late toxicity RT related | from January 2010 to December 2023
  Evaluation of toxicities related to radiotherapy treatment using the scale CTCAE (Grade 1: Mild, Grade 2: Moderate, Grade 3: Severe, Grade 4: Life-threatening, Grade 5: Death)

CONTACTS AND LOCATIONS:
Locations (28):
- Italy (28):
  - Aorn San Pio, Benevento, Benevento
  - Humanitas Gavazzeni, Bergamo, Bergamo
  - Ospedale Perrino, Brindisi, BR
  - Spedali Civili, Brescia, BS
  - Responsible Research Hospital, Campobasso, CB
  - Azienda Ospedaliera Universitaria Careggi, Florence, Firenze
  - Irccs Ospedale Policlinico San Martino, Genova, Genova
  - A.O.U. "G. Martino" - Università degli Studi di Messina, Messina, Messina
  - Fondazione I.R.C.C.S Istituto Nazionale Tumori di Milano, Milan, MILANO
  - IEO, Milan, Milano
  - IRCCS Humanitas Research Humanitas, Rozzano, MILANO
  - IRCCS Ospedale San Raffaele, Milan, Milan
  - INT IRCCS Fondazione G. Pascale, Napoli, Napoli
  - Ospedale Maggiore della Carita, Novara, NOVARA
  - Civico Palermo, Palermo, Palermo
  - Istituto Oncologico Veneto, Padua, PD
  - Azienda Ospedaliera Universitaria Pisana, Pisa, PI
  - IRCCS Centro di Riferimento Oncologico di Aviano, Aviano, Pordenone
  - Uo Radioterapia Aor San Carlo, Potenza, PZ
  - Irccs Crob, Rionero in Vulture, PZ
  - UOC Radioterapia Ospedale San Filippo Neri, Roma, RM
  - Azienda Ospedaliera San Giovanni Addolorata, Roma, RM
  - Fondazione Policlinico Universitario, Campus-Biomedico, Roma, Roma
  - Fondazione PTV Policlinico Tor Vergata, Roma, Roma
  - Azienda Ospedaliera Sant'Andrea, Roma, Roma
  - S.C. Radioterapia Oncologica ASL Taranto, Taranto, Taranto
  - Radioterapia Oncologica - Ospedale Sanata Chiara, Trento, TRENTO
  - S.C. Radioterapia Oncologica - Azienda Ospedaliera Santa Maria Terni, Terni, TR

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] T. G. S. L. C. M. V. M.-J. T. V. P. T. G. W. G. S. S. Annemiek van Ommen-Nijhof, "Survival and prognostic factors in oligometastatic breast cancer," the breast, 2022.
- [Background] K. A. W. W. A. W. V. F. B. J. K. Steven J. Chmura, "NRG-BR002: A phase IIR/III trial of standard of care systemic therapy with or without stereotactic body radiotherapy (SBRT) and/or surgical resection (SR) for newly oligometastatic breast cancer," ASCO, 2022
- [Background] D. A. P. Stephen Harrow, "Stereotactic Radiation for the Comprehensive Treatment of Oligometastases (SABR-COMET) - Extended Long-Term Outcomes," International Journal of Radiation Oncology, Biology, Physics, 2022.
- [Background] N. N. Terao M, "Diagnosis of oligometastasis," Transl Cancer Res., 2020